CLINICAL TRIAL: NCT07322237
Title: Empagliflozin + Carvedilol vs. Carvedilol Alone for Patients With Cirrhosis and Left Ventricular Diastolic Dysfunction and Impact on Hepatic Decompensation and Survival: A Double-Blind Placebo-Controlled Randomized Controlled Trial
Brief Title: DICE Study- Diastolic Improvement With Carvedilol & Empagliflozin in Patients With Cirrhosis
Acronym: DICE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Madhumita Premkumar, Additional Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PGI/IEC/2025/SPL-865
Record Dates: First submitted 2025-11-30; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Cirrhotic Cardiomyopathy; Empagliflozin; Cardiometabolic Risk Factors; Cirrhosis
Keywords: Empagliflozin in cirrhosis; Carvedilol in Cirrhosis; SGLT-2 inhibitor; Ascites; Diastolic heart failure; heart failure with preserved ejection fraction
MeSH Terms: conditions — Fibrosis; Ascites; Heart Failure, Diastolic | interventions — empagliflozin; Carvedilol

STUDY DESIGN:
Intervention Model Description: Double Blind Placebo controlled Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Empagliflozin + Carvedilol-arm (Active Comparator): Experimental: Empagliflozin + Carvedilol-arm
  * Empagliflozin fixed dose of 10 mg per day in patients with or without diabetes for 1 year from randomization
  * Carvedilol: Starting dose of 3.125 mg twice daily targeted upwards q 7 days to achieve target heart rate
  * Standard Medical Therapy for liver disease as per clinician decision
  Interventions: Drug: Empagliflozin + Carvedilol
- Active Comparator: Carvedilol arm (Active Comparator): * Carvedilol: Starting dose of 3.125 mg twice daily targeted upwards q 7 days to achieve target heart rate 10 mg placebo administered once daily.
  * Standard Medical Therapy prescribed as per clinician decision
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Empagliflozin + Carvedilol — Patient Recruitment:
  The study participants are all cirrhosis patients receiving treatment at PGIMER Chandigarh. Eligible participants meeting LVDD criteria per the CCM Consortium 2020 consensus.
  Carvedilol Dosing protocol in this study Patients will be given carvedilol in a starting dose of 3.125 mg twice daily. The dose will be titrated weekly to achieve a target heart rate of 50-60/ min taking care that side effects such as hypotension bronchospasm excessive bradycardia are not seen. The maximum dosage allowed as per prior trial data is 25 mg per day.
  Empagliflozin Dosing protocol in this Study:
  • All patients will receive a standard dose of Empagliflozin fixed dose of 10 mg per day in patients with or without diabetes.
  Arms: Experimental: Empagliflozin + Carvedilol-arm
Drug: Carvedilol — * Carvedilol: Starting dose of 3.125 mg twice daily targeted upwards q 7 days to achieve target heart rate 10 mg placebo pill
  * Standard Medical Therapy
  Arms: Active Comparator: Carvedilol arm

SUMMARY:
1. This proposed double-blind placebo controlled randomized controlled trial incorporates recent advances in management of heart failure and portal hypertension using the SGLT-2 inhibitor i.e. EMPAGLIFLOZIN. The drug has been found to be useful in large trials on heart failure with preserved ejection fraction in the general population with improvement in MASLD progression, with improvement in body weight and hepatic steatosis but no change in liver fibrosis.
2. Sodium-glucose cotransporter 2 (SGLT2) inhibitors have been shown to reduce the development and progression of heart failure in patients with type 2 diabetes and in those with heart failure and a reduced and preserved ejection fraction. In patients with cirrhosis safety of empagliflozin in a dose of 10 mg has been demonstrated.
3. Prevention of decompensation related events in cirrhosis is the key endpoint of any liver-directed therapy as the median survival in the compensated state exceeds 10 years but median survival in the decompensated state approximates 1.5 years. Previous data has demonstrated the risk of hepatic decompensation acute kidney injury and poor survival in patients with cirrhosis and heart failure with preserved ejection fraction (HFpEF) i.e. LVDD a large subset of whom meet criteria for CCM.

DETAILED DESCRIPTION:
New diagnostic criteria for cirrhotic cardiomyopathy For the diagnosis of cirrhotic cardiomyopathy (CCM) we will use criteria proposed by the CCM consortium in 2020 with modification to take septal e' and E/e' readings. In accordance with the recent CCM criteria 'systolic dysfunction is defined as an ejection fraction (EF) of 50% or less or an absolute value of GLS <18%. LVDD grade will be determined if 3 of the following 4 criteria are met: early diastolic trans mitral flow to early diastolic mitral annular velocity (E/e') ≥15 left atrial volume index (LAVI) >34 mL/m2 septal early diastolic mitral annular velocity (e') <7 cm/second or tricuspid regurgitation (TR) maximum velocity >2.8 m/second in the absence of pulmonary hypertension (HTN) and the presence of measurable early to late diastolic trans mitral flow velocity (E/A) ratio (E/A >2 = grade 3 E/A 0.8-2 = grade 2)'. LVDD will be classified as "of indeterminate grade" when only 2 of the 4 criteria are met. The supporting criteria for diagnosis of LVDD are changes in cardiac chamber sizes electrophysiological abnormalities increased biomarkers like N terminal pro-brain natriuretic peptide (NT-Pro BNP) and troponin I.

ELIGIBILITY:
Inclusion criteria

* Age range of 18-65 years
* Cirrhosis as diagnosed by histology or clinical laboratory and USG findings
* LVDD (with EF>50%) on 2D echocardiography with TDI
* Written informed consent.

Exclusion criteria

* Age >65 years
* Serum Creatinine>2 mg/dl
* History of urinary tract /genital infections in last 3 months
* Patient on treatment with statin (one month before the study)
* Advanced Cirrhosis (MELD>20)
* Coronary artery disease
* Sick sinus syndrome/ Pacemaker valvular heart disease
* Cardiac rhythm disorder Peripartum cardiomyopathy
* Portopulmonary hypertension/ hepatopulmonary syndrome
* Transjugular intrahepatic porto systemic shunt (TIPS) insertion
* Hepatocellular carcinoma
* Pregnancy or lactation
* Patients with HIV or retroviral therapy
* Anemia Hb < 8gm/dl in females and < 9 gm/dl in males
* Acute variceal bleeding in last 6months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-01-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite end point of decompensation event and/or death | From enrolment through study completion, an average of 1 year
  The primary outcome measure is defined as a composite end point of acute decompensation event (acute variceal bleeding new ascites or recurrence of previously controlled ascites episode of hepatic encephalopathy or acute kidney injury) OR all-cause death in patients with cirrhosis and LVDD

SECONDARY OUTCOMES:
Improvement in Cardiac Diastolic Function | From enrolment through study completion, an average of 1 year
  Improvement in CCM parameters (left ventricular diastolic function) in either arm based on Echocardiography and Cardiac Imaging
  Septal E/e' ratio
Improvement in Cardiac Diastolic Function | From enrolment through study completion, an average of 1 year
  Improvement in CCM parameters (left ventricular diastolic function) in either arm based on Echocardiography and Cardiac Imaging Septal e' velocity
Improvement in Cardiac Diastolic Function | From enrolment through study completion, an average of 1 year
  Improvement in CCM parameters (left ventricular diastolic function) in either arm based on Echocardiography and Cardiac Imaging
  Left atrial volume index
Improvement in Cardiac Diastolic Function | From enrolment through study completion, an average of 1 year
  Improvement in CCM parameters (left ventricular diastolic function) in either arm based on Echocardiography and Cardiac Imaging
  Tricuspid regurgitant Velocity
Improvement in Cardiac Systolic Function | From enrolment through study completion, an average of 1 year
  Improvement in Cardiac systolic function (Cardiac Index) in either arm based on Echocardiography and Cardiac Imaging
Improvement in Cardiac Systolic Function | From enrolment through study completion, an average of 1 year
  Improvement in Cardiac systolic function (Ejection Fraction) in either arm based on Echocardiography and Cardiac Imaging
Improvement in Cardiac Systolic Function | From enrolment through study completion, an average of 1 year
  Improvement in Cardiac systolic function (Global Longitudinal Strain) in either arm based on Echocardiography and Cardiac Imaging
Hospitalization events | From enrolment through study completion, an average of 1 year
  • Episodes warranting hospitalization
• Serum level of NT-proBNP | At enrolment
  Cardiac biomarkers
• Serum level of NT-proBNP | At 6 months from enrolment
  Cardiac biomarkers
• Serum level of NT-proBNP | At 12 months from enrolment
  Cardiac biomarkers
• Serum level of Galectin-3 | At enrolment
  Cardiac biomarkers
• Serum level of Galectin 3 | At 6 months from enrolment
  Cardiac biomarkers
• Serum level of Galectin 3 | At 12 months from enrolment
  Cardiac biomarkers
• Serum level of Aldosterone | At enrolment
  Cardiac biomarkers
• Serum level of Aldosterone | At 6 months from enrolment
  Cardiac biomarkers- Renin angiotensin aldosterone system
• Serum level of Aldosterone | At 12 months from enrolment
  Cardiac biomarkers- Renin angiotensin aldosterone system

CONTACTS AND LOCATIONS:
Locations (1):
- PGIMER Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No
This database has identifier information